CLINICAL TRIAL: NCT02366819
Title: PERIOP-FOLFIRINOX: A Pilot Trial of Perioperative Genotype-guided Irinotecan Dosing of gFOLFIRINOX for Locally Advanced Gastroesophageal Adenocarcinoma
Brief Title: Genetic Analysis-Guided Irinotecan Hydrochloride Dosing of mFOLFIRINOX in Treating Patients With Locally Advanced Gastroesophageal or Stomach Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-0594; NCI-2014-02574 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB14-0594 (Other: University of Chicago); P30CA014599 (NIH)
Record Dates: First submitted 2015-01-27; First posted 2015-02-19 (Estimated); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Adenocarcinoma; Gastric Adenocarcinoma; Stage IIB Gastric Cancer; Stage IIIA Esophageal Adenocarcinoma; Stage IIIA Gastric Cancer; Stage IIIB Esophageal Adenocarcinoma; Stage IIIB Gastric Cancer; Stage IIIC Esophageal Adenocarcinoma; Stage IIIC Gastric Cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Stomach Neoplasms | interventions — Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil; Surgical Procedures, Operative; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (mFOLFIRINOX, surgery) (Experimental): PREOPERATIVE THERAPY: Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and fluorouracil IV over 46 hours continuously on day 1. Courses repeat every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  SURGERY: Patients undergo conventional surgery.
  POST-OPERATIVE THERAPY: Beginning 5-10 weeks after surgery, patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and fluorouracil IV over 46 hours continuously on day 1. Courses repeat every 2 weeks for 4 more courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin Calcium; Drug: Irinotecan Hydrochloride; Drug: Fluorouracil; Procedure: Conventional Surgery

INTERVENTIONS:
Drug: Oxaliplatin — Given IV
Drug: Leucovorin Calcium — Given IV
  Other Names: CF
Drug: Irinotecan Hydrochloride — Given IV
Drug: Fluorouracil — Given IV
Procedure: Conventional Surgery — Undergo surgery
  Other Names: surgery, conventional

SUMMARY:
This pilot clinical trial studies genetic analysis-guided irontecan hydrochloride dosing of modified fluorouracil, irinotecan hydrochloride, leucovorin calcium, oxaliplatin (mFOLFIRINOX) in treating patients with gastroesophageal or stomach cancer that has spread from where it started to nearby tissue or lymph nodes. Drugs used in chemotherapy, such as fluorouracil, irinotecan hydrochloride, leucovorin calcium, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Leucovorin calcium may also help fluorouracil work better. Genetic analysis may help doctors determine what dose of irinotecan hydrochloride patients can tolerate.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the residual tumor (R) 0 resection rate. II. To determine the pathologic complete response (pCR) rate of up to 36 patients treated with 4 cycles of neoadjuvant mFOLFIRINOX (UGTA1A1 genotype-dosed irinotecan [irinotecan hydrochloride]) regimen.

SECONDARY OBJECTIVES:

I. Response rate (radiographic [computed tomography (CT)], and metabolic (positron emission tomography [PET] maximum standardized uptake value [SUVmax]) to chemotherapy.

II. Chemotherapy-related toxicity. III. Surgical morbidity. IV. Overall survival (OS) measured from the time of histologic diagnosis. V. Disease-free survival measured from the time of histologic diagnosis. VI. Pattern of recurrence (distant, locoregional, both). VII. Human epidermal growth factor receptor 2 positive (HER2+) vs HER2 negative (-) difference in clinical outcomes.

OUTLINE:

PREOPERATIVE THERAPY: Patients receive oxaliplatin intravenously (IV) over 2 hours, leucovorin calcium IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and fluorouracil IV over 46 hours continuously on day 1. Courses repeat every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

SURGERY: Patients undergo surgery.

POST-OPERATIVE THERAPY: Beginning 5-10 weeks after surgery, patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and fluorouracil IV over 46 hours continuously on day 1. Courses repeat every 2 weeks for 4 more courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced gastric (primary endpoint includes proximal and mid-body stomach) or esophagogastric adenocarcinoma; distal gastric (antral) adenocarcinomas are eligible for enrolment but will not be included in the primary analysis
* Locally advanced disease as determined by endoscopic ultrasound (EUS) stage > primary tumor (T) 3 and/or any T, lymph nodes (N)+ disease without metastatic disease (Mx)
* All patients must have diagnostic laparoscopy with diagnostic washings for cytology; both cytology positive and negative patients are eligible for enrolment, but only cytology negative patients will be included in the primary analyses; gross peritoneal disease is not eligible
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Eligible for surgery with curative intent
* Absolute neutrophil count (ANC) >= 1250/ul
* Hemoglobin >= 9 g/dL
* Platelets >= 100,000/ul
* Total bilirubin < 1.5 x upper limit of normal
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) < 2.5 x upper limit of normal for patients without liver metastases OR SGOT and SGPT < 5 x upper limit of normal for patients with liver metastases
* Creatinine =< 1.5 x upper limit of normal
* Measurable or non-measurable disease by Response Evaluation Criteria in Solid Tumor (RECIST) 1.1 will be allowed
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, up until 30 days after final study treatment; should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients taking substrates, inhibitors, or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) should be encouraged to switch to alternative drugs whenever possible, given the potential for drug-drug interactions with irinotecan
* Signed informed consent

Exclusion Criteria:

* Previous or concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or any other cancer for which the patient has been previously treated and the lifetime recurrence risk is less than 30%
* Inflammatory bowel disease that is uncontrolled or on active treatment (Crohn's disease, ulcerative colitis)
* Diarrhea, grade 1 or greater by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, version [v] 4.0)
* Neuropathy, grade 2 or greater by NCI-CTCAE, v 4.0
* Serious underlying medical or psychiatric illnesses that would, in the opinion of the treating physician, substantially increase the risk for complications related to treatment
* Active uncontrolled bleeding
* Pregnancy or breastfeeding
* Major surgery within 4 weeks
* Patients with any polymorphism in UGT1A1 other than *1 or *28 (e.g, *6) will be allowed and treated as in the *28/*28 dosing group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-12-11 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
R0 (analysis will be performed evaluating the R0 rate) | During surgery
  Intention-to-treat analysis will be performed, and patients with tumor progression during/after neoadjuvant chemotherapy that precludes surgery will be included as non-R0 resection. A subset analysis will be performed evaluating the R0 rate for those patients actually undergoing surgery.

SECONDARY OUTCOMES:
Response rate | Up to 5 years
  Will be evaluated by reporting event rates along with exact (binomial distribution-based) 95% confidence intervals.
Surgical morbidity | Up to 5 years
  Will be evaluated by reporting event rates along with exact (binomial distribution-based) 95% confidence intervals.
Pattern of recurrence | Up to 5 years
  Will be evaluated by reporting event rates along with exact (binomial distribution-based) 95% confidence intervals.
Incidence of toxicity based on NCI-CTCAE v 4.0 | Up to 5 years
  Toxicities will be summarized by type, grade, and attribution.
OS (estimated using the Kaplan-Meier procedure and compared in the subgroups of patients with and without pCR (grade 1a) using the log-rank test) | Time from enrollment/registration to the time of death, of any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier procedure and compared in the subgroups of patients with and without pCR (grade 1a) using the log-rank test.
Progression free survival | Time from enrollment/registration to time of progression or death from any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier procedure and compared in the subgroups of patients with and without pCR (grade 1a) using the log-rank test.

OTHER OUTCOMES:
Circulating tumor cell (CTC) numbers derived from portal and peripheral blood samples | Up to 5 years
  Pearson or Spearman rank correlation coefficients will be calculated between CTC numbers derived from portal and peripheral blood samples.
Change in SUVmax for PET/CT studies | Baseline to after 8 weeks of chemotherapy
  Will be analyzed lesion-by-lesion using paired t-tests or Wilcoxon, signed rank tests.
Change in SUVmax for the primary esophageal tumor | Baseline to up to 5 years
  Will be correlated with clinical and histopathological response rates by logistic regression, and with progression-free and overall survival by Cox regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Catenacci, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Kellogg Cancer Center - Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois

REFERENCES:
- [Derived] Catenacci DVT, Chase L, Lomnicki S, Karrison T, de Wilton Marsh R, Rampurwala MM, Narula S, Alpert L, Setia N, Xiao SY, Hart J, Siddiqui UD, Peterson B, Moore K, Kipping-Johnson K, Markevicius U, Gordon B, Allen K, Racette C, Maron SB, Liao CY, Polite BN, Kindler HL, Turaga K, Prachand VN, Roggin KK, Ferguson MK, Posner MC. Evaluation of the Association of Perioperative UGT1A1 Genotype-Dosed gFOLFIRINOX With Margin-Negative Resection Rates and Pathologic Response Grades Among Patients With Locally Advanced Gastroesophageal Adenocarcinoma: A Phase 2 Clinical Trial. JAMA Netw Open. 2020 Feb 5;3(2):e1921290. doi: 10.1001/jamanetworkopen.2019.21290. PMID 32058557